CLINICAL TRIAL: NCT01368393
Title: Electroacupuncture Analgesia for Colonoscopy: a Prospective, Randomized, Double-blind, Sham-controlled Study
Brief Title: Electroacupuncture Analgesia for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2010.404
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (Experimental)
  Interventions: Procedure: Electroacupuncture
- Sham acupuncture (Active Comparator)
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Patients randomized to the experimental group will receive electroacupuncture at acupoints relevant to the treatment of abdominal pain and anxiety, including Zusanli (stomach meridian ST-36), Hegu (large intestine meridian LI-4), and Neiguan (pericardium meridian PC-6). Electric stimulation will be employed to the needles
  Arms: Electroacupuncture
Procedure: Sham acupuncture — Sterile blunt-tip needles will be placed (without skin penetration) 15 mm away from the acupoints. "Pseudostimulation" will be given by deliberately connecting the needle to the incorrect output socket of the electroacupuncture device, thus there will be no flow of electric current.
  Arms: Sham acupuncture

SUMMARY:
Background:

Colonoscopy is often regarded as a painful and unpleasant procedure. Electroacupuncture (EA) has been used successfully to treat pain of various origins, but few good-quality studies have evaluated its role in treating pain and anxiety during colonoscopy.

Objective:

To investigate the efficacy of EA in reducing procedure-related pain and the consumption of sedatives/analgesics during colonoscopy.

Design:

Prospective, randomized, double-blind, sham-controlled study.

Subjects:

One hundred and twenty eight consecutive patients undergoing first-time elective day-case colonoscopy without previous experience of acupuncture will be recruited.

Interventions:

Patients will be randomized to receive either 45 minutes of EA or sham acupuncture (SA) before colonoscopy. The acupoints relevant to the treatment of abdominal pain, including Zusanli, Hegu, and Neiguan will be used. For the SA group, blunt-tip needles will be placed (without skin penetration) 15 mm away from the acupoints. Foam blocks will be used to stabilize the needles and to blind the patients and endoscopists to the treatment allocation. EA and SA will be continued throughout colonoscopy. A mixture of Propofol and Alfentanil, delivered by a patient-controlled syringe pump, will be used for sedation/analgesia in both groups.

Outcome measures:

Primary outcome: doses of patient-controlled sedation/analgesia consumed. Secondary outcomes: pain and satisfaction scores according to a visual analog scale, cecal intubation rate/time, and episodes of hypotension/desaturation.

ELIGIBILITY:
Inclusion criteria:

* Consecutive patients (aged between 18 and 60 years) undergoing first-time elective day-case colonoscopy
* Patients with American Society of Anesthesiologists (ASA) grading I-II
* Informed consent available

Exclusion criteria:

* Patients with previous experience of acupuncture
* Patients with previous history of colorectal surgery
* Patients who are diagnosed with irritable bowel syndrome according to Rome III criteria
* Patients with chronic pain syndrome
* Patients with psychiatric disorder
* Patients with poor cognitive function
* Patients with renal impairment
* Patients with obstructive sleep apnea syndrome
* Patients with cardiac arrhythmias
* Patients with cardiac pacemaker
* Patients who are pregnant
* Patients who are allergic to the acupuncture needles or Propofol/Alfentanil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Dose of patient-controlled sedation/analgesia consumed | During the procedure (up to 1 day)

SECONDARY OUTCOMES:
Pain score | During the procedure (up to 1 day)
  Using a 10-cm unscaled visual analog scale; 0 = no pain, 10 = very painful
Patients' satisfaction score | During the procedure (up to 1 day)
  Using a 10-cm unscaled visual analog scale; 0 = not satisfied, 10 = very satisfied
Patients' willingness to repeat the procedure | Up to 1 day
Endoscopists' satisfaction score | During the procedure (up to 1 day)
  Using a 10-cm unscaled visual analog scale; 0 = not satisfied, 10 = very satisfied
Cecal intubation rate | During the procedure (up to 1 day)
  Complete colonoscopy is defined as identification of ileocecal valve
Cecal intubation time | During the procedure (up to 1 day)
  The time from introduction of the colonoscope to the cecum
Total procedure time | During the procedure (up to 1 day)
Episodes of hypotension | During the procedure (up to 1 day)
  Defined as systolic blood pressure <90 mmHg
Episodes of desaturation | During the procedure (up to 1 day)
  Defined as SaO2 <90%

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong SAR, China